CLINICAL TRIAL: NCT01844661
Title: Phase 1 Trial of Celyvir in Children and Adults With Metastatic and Refractory Solid Tumors.
Brief Title: Safety and Efficacy of Repeated Infusion of CELYVIR in Children and Adults With Metastatic and Refractory Tumors.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Manuel Ramírez, MD PhD, Dr., Hospital Infantil Universitario Niño Jesús, Madrid, Spain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT2008-000364-16
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Children; Solid Tumors; Metastases
Keywords: Mesenchymal stem cells; Oncolytic adenovirus
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CELYVIR (Experimental): Patients will received weekly (n=6) IV infusion of Celyvir.
  Interventions: Biological: CELYVIR

INTERVENTIONS:
Biological: CELYVIR
  Other Names: Bone marrow-derived autologous mesenchymal stem cells infected with ICOVIR5, an oncolytic adenovirus.

SUMMARY:
The investigators will evaluate the safety of weekly infusions (n=6) of CELYVIR in children and adults with metastatic and refractory solid tumors. CELYVIR consists in bone marrow-derived autologous mesenchymal stem cells (MSCs) infected with ICOVIR5, an oncolytic adenovirus. In addition to data on toxicities the investigators will evaluate clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Children: Up to 18 yrs. Refractory to at least 2 previous therapy lines. Life expectancy more than 6 months. Measurable disease.
* Adults: 18-75 yrs. Refractory to at least 2 previous therapy lines. ECOG (Eastern Cooperative Oncology Group) <2. Measurable disease.

Exclusion Criteria:

* Pregnancy.
* Central Nervous System metastasis.
* Experimental therapy during the previous month.
* Chemotherapy less than 3 weeks previous.
* Any organ functionally impaired.
* Concurrent infectious disease.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Adverse effects after intravenous infusions | 48 hours after each infusion
  We will record any sign or symptom that could be related to the infusion of Celyvir.

SECONDARY OUTCOMES:
Clinical outcome | Up to 2 months after the last infusion
  Clinical outcome will be labelled as complete response, partial response, stable disease or disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Ramírez, MD PhD, Principal Investigator — Hospital Universitario Niño Jesús
Locations (1):
- Hospital Universitario Niño Jesús, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Morales-Molina A, Gambera S, Leo A, Garcia-Castro J. Combination immunotherapy using G-CSF and oncolytic virotherapy reduces tumor growth in osteosarcoma. J Immunother Cancer. 2021 Mar;9(3):e001703. doi: 10.1136/jitc-2020-001703. PMID 33737338
- [Derived] Ruano D, Lopez-Martin JA, Moreno L, Lassaletta A, Bautista F, Andion M, Hernandez C, Gonzalez-Murillo A, Melen G, Alemany R, Madero L, Garcia-Castro J, Ramirez M. First-in-Human, First-in-Child Trial of Autologous MSCs Carrying the Oncolytic Virus Icovir-5 in Patients with Advanced Tumors. Mol Ther. 2020 Apr 8;28(4):1033-1042. doi: 10.1016/j.ymthe.2020.01.019. Epub 2020 Jan 21. PMID 32053771